CLINICAL TRIAL: NCT01129596
Title: Post-marketing Surveillance of Long-term Administration of Donepezil Hydrochloride -Investigation of the Clinical Condition and Safety in Patients With Alzheimer's Disease-
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: ART05T
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: donepezil hydrochloride

INTERVENTIONS:
Drug: donepezil hydrochloride — This is a multicenter, open-labeled, practice-based, post-marketing surveillance study. Therefore, dosing is not specified.

SUMMARY:
The purpose of this study is to investigate the following about donepezil hydrochloride administration in patients with mild or moderate Alzheimer's Disease in clinical practice: cognitive function, Functional Assessment Staging (FAST) score, adverse events/adverse drug reactions, and patient background.

ELIGIBILITY:
Inclusion criteria:

Patients diagnosed with Alzheimer's Disease by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Patients diagnosed with mild or moderate Alzheimer's Disease, applicable to FAST score 4 or 5.

Exclusion criteria:

Patients with history of hypersensitivity to component of Aricept or piperidine derivative. Patients registered for this survey before.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital, Clinical. Japan
Sampling Method: Non-Probability Sample
Enrollment: 10238 (Actual)
Dates: Start 2010-06-10 (Actual); Primary Completion 2015-09-25 (Actual); Study Completion 2016-06-23 (Actual)

PRIMARY OUTCOMES:
The transition of clinical condition is evaluated comparing the result of HDS-R,MMSE with the time of study initiation | 48 months(12 weeks and every 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Kenta Sumitomo, Study Director — Drug Fostering and Evolution Coordination Department, Eisai Co., Ltd.
Locations (722):
- Japan (722):
  - Aisai, Aichi-ken
  - Chita, Aichi-ken
  - Gamagōri, Aichi-ken
  - Handa, Aichi-ken
  - Ichinomiya, Aichi-ken
  - Inazawa, Aichi-ken
  - Inuyama, Aichi-ken
  - Kariya, Aichi-ken
  - Kasugai, Aichi-ken
  - Komaki, Aichi-ken
  - Kōnan, Aichi-ken
  - Nagoya, Aichi-ken
  - Nishio, Aichi-ken
  - Nisshin, Aichi-ken
  - Okazaki, Aichi-ken
  - Owariasahi, Aichi-ken
  - Ōbu, Aichi-ken
  - Seto, Aichi-ken
  - Shinshiro, Aichi-ken
  - Tahara, Aichi-ken
  - Tokoname, Aichi-ken
  - Toyoake, Aichi-ken
  - Toyohashi, Aichi-ken
  - Toyokawa, Aichi-ken
  - Toyota, Aichi-ken
  - Tōkai, Aichi-ken
  - Yatomi, Aichi-ken
  - Daisen, Akita
  - Katagami, Akita
  - Oga, Akita
  - Ōdate, Akita
  - Semboku, Akita
  - Yokote, Akita
  - Yurihonjō, Akita
  - Yuzawa, Akita
  - Goshogawara, Aomori
  - Hachinohe, Aomori
  - Hirosaki, Aomori
  - Kamikita, Aomori
  - Kitatsugaru, Aomori
  - Mutsu, Aomori
  - Sannohe, Aomori
  - Towada, Aomori
  - Abiko, Chiba
  - Asahi, Chiba
  - Choshi, Chiba
  - Funabashi, Chiba
  - Ichihara, Chiba
  - Ichikawa, Chiba
  - Inzai, Chiba
  - Isumi, Chiba
  - Kashiwa, Chiba
  - Katori-shi, Chiba
  - Kimitsu, Chiba
  - Kisarazu, Chiba
  - Matsudo, Chiba
  - Mobara, Chiba
  - Nagareyama, Chiba
  - Narita, Chiba
  - Sakura, Chiba
  - Sambu, Chiba
  - Sanmu, Chiba
  - Tateyama, Chiba
  - Tōgane, Chiba
  - Yachimata, Chiba
  - Yachiyo, Chiba
  - Yotsukaidō, Chiba
  - Imabari, Ehime
  - Iyo, Ehime
  - Kamiukena, Ehime
  - Matsuyama, Ehime
  - Minamiuwa, Ehime
  - Niihama, Ehime
  - Ōzu, Ehime
  - Saijō, Ehime
  - Seiyo, Ehime
  - Shikokuchūō, Ehime
  - Tōon, Ehime
  - Uwajima, Ehime
  - Yawatahama, Ehime
  - Echizen, Fukui
  - Katsuyama, Fukui
  - Mikatakaminaka, Fukui
  - Obama, Fukui
  - Sabae, Fukui
  - Sakai, Fukui
  - Tsuruga, Fukui
  - Asakura, Fukuoka
  - Chikugo, Fukuoka
  - Chikushi, Fukuoka
  - Chikushino-shi, Fukuoka
  - Fukutsu, Fukuoka
  - Iizuka, Fukuoka
  - Itoshima, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Kurume, Fukuoka
  - Miyako, Fukuoka
  - Miyama, Fukuoka
  - Nakama, Fukuoka
  - Nōgata, Fukuoka
  - Ogōri, Fukuoka
  - Omuta, Fukuoka
  - Ōnojō, Fukuoka
  - Tagawa, Fukuoka
  - Ukiha, Fukuoka
  - Wakasugi, Fukuoka
  - Yanagawa, Fukuoka
  - Yukuhashi, Fukuoka
  - Aizu-Wakamatsu, Fukushima
  - Date, Fukushima
  - Futaba, Fukushima
  - Higashishirakawa, Fukushima
  - Ishikawa, Fukushima
  - Iwaki, Fukushima
  - Kitakata, Fukushima
  - Kōriyama, Fukushima
  - Nihommatsu, Fukushima
  - Onuma, Fukushima
  - Sōma, Fukushima
  - Sukagawa, Fukushima
  - Tamura, Fukushima
  - Yama, Fukushima
  - Ena, Gifu
  - Gujō, Gifu
  - Hashima, Gifu
  - Minokamo, Gifu
  - Mizuho, Gifu
  - Nakatsugawa, Gifu
  - Ōgaki, Gifu
  - Sekimachi, Gifu
  - Tajimi, Gifu
  - Takayama, Gifu
  - Toki, Gifu
  - Yamagata, Gifu
  - Fujioka, Gunma
  - Isesaki, Gunma
  - Kiryū, Gunma
  - Kitagumma, Gunma
  - Maebashi, Gunma
  - Numata, Gunma
  - Ōta, Gunma
  - Ōwa, Gunma
  - Shibukawa, Gunma
  - Takasaki, Gunma
  - Tatebayashi, Gunma
  - Tomioka, Gunma
  - Tone, Gunma
  - Aki, Hiroshima
  - Fuchū, Hiroshima
  - Fukuyama, Hiroshima
  - Higashihiroshima, Hiroshima
  - Kure, Hiroshima
  - Mihara, Hiroshima
  - Miyoshi, Hiroshima
  - Onomichi, Hiroshima
  - Ōtake, Hiroshima
  - Shōbara, Hiroshima
  - Takehara, Hiroshima
  - Abashiri, Hokkaido
  - Akkeshi, Hokkaido
  - Asahikawa, Hokkaido
  - Ashibetsu, Hokkaido
  - Bibai, Hokkaido
  - Chitose, Hokkaido
  - Date, Hokkaido
  - Ebetsu, Hokkaido
  - Eniwa, Hokkaido
  - Fukagawa, Hokkaido
  - Furano, Hokkaido
  - Hakodate, Hokkaido
  - Hiroo, Hokkaido
  - Hokuto, Hokkaido
  - Ishikari, Hokkaido
  - Iwamizawa, Hokkaido
  - Kameda, Hokkaido
  - Kamikawa, Hokkaido
  - Kato, Hokkaido
  - Kawakami, Hokkaido
  - Kitami, Hokkaido
  - Kushiro, Hokkaido
  - Mombetsu, Hokkaido
  - Muroran, Hokkaido
  - Nakagawa, Hokkaido
  - Nayoro, Hokkaido
  - Noboribetsu, Hokkaido
  - Obihiro, Hokkaido
  - Otaru, Hokkaido
  - Rumoi, Hokkaido
  - Sapporo, Hokkaido
  - Shibetsu, Hokkaido
  - Sorachi, Hokkaido
  - Sōya, Hokkaido
  - Sunagawa, Hokkaido
  - Tomakomai, Hokkaido
  - Yoichi, Hokkaido
  - Yūfutsu, Hokkaido
  - Akashi, Hyōgo
  - Ako, Hyōgo
  - Amagasaki, Hyōgo
  - Asago, Hyōgo
  - Ashiya, Hyōgo
  - Awaji, Hyōgo
  - Himeji, Hyōgo
  - Itami, Hyōgo
  - Kakogawa, Hyōgo
  - Kako, Hyōgo
  - Kasai, Hyōgo
  - Katō, Hyōgo
  - Kawabe, Hyōgo
  - Kawanishi, Hyōgo
  - Kobe, Hyōgo
  - Miki, Hyōgo
  - Nishinomiya, Hyōgo
  - Sanda, Hyōgo
  - Shisō, Hyōgo
  - Sumoto, Hyōgo
  - Takarazuka, Hyōgo
  - Takasago, Hyōgo
  - Tamba, Hyōgo
  - Tatsuno, Hyōgo
  - Toyooka, Hyōgo
  - Yabu, Hyōgo
  - Bandō, Ibaraki
  - Chikusei, Ibaraki
  - Higashiibaraki, Ibaraki
  - Hitachi, Ibaraki
  - Hitachi-Naka, Ibaraki
  - Hitachiota, Ibaraki
  - Inashiki, Ibaraki
  - Ishioka, Ibaraki
  - Jōsō, Ibaraki
  - Kamisu, Ibaraki
  - Kasama, Ibaraki
  - Koga, Ibaraki
  - Mito, Ibaraki
  - Moriya, Ibaraki
  - Naka, Ibaraki
  - Ryūgasaki, Ibaraki
  - Sashima, Ibaraki
  - Takahagi, Ibaraki
  - Toride, Ibaraki
  - Tsuchiura, Ibaraki
  - Tsukuba, Ibaraki
  - Tsukubamirai, Ibaraki
  - Ushiku, Ibaraki
  - Yūki, Ibaraki
  - Hakusan, Ishikawa-ken
  - Kahoku, Ishikawa-ken
  - Kanazawa, Ishikawa-ken
  - Komatsu, Ishikawa-ken
  - Nanao, Ishikawa-ken
  - Suzu, Ishikawa-ken
  - Wajima, Ishikawa-ken
  - Hanamaki, Iwate
  - Ichinoseki, Iwate
  - Kamaishi, Iwate
  - Kitakami, Iwate
  - Miyako, Iwate
  - Morioka, Iwate
  - Ninohe, Iwate
  - Numakunai, Iwate
  - Ōshū, Iwate
  - Tōno, Iwate
  - Ayauta, Kagawa-ken
  - Kan’onjichō, Kagawa-ken
  - Kita, Kagawa-ken
  - Marugame, Kagawa-ken
  - Mitoyo, Kagawa-ken
  - Sakaidechō, Kagawa-ken
  - Sanuki, Kagawa-ken
  - Shozu, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Aira, Kagoshima-ken
  - Amami, Kagoshima-ken
  - Hioki, Kagoshima-ken
  - Ibusuki, Kagoshima-ken
  - Ichikikushikino, Kagoshima-ken
  - Izumi, Kagoshima-ken
  - Kanoya, Kagoshima-ken
  - Kirishima, Kagoshima-ken
  - Makurazaki, Kagoshima-ken
  - Minamikyushu, Kagoshima-ken
  - Nishinomote, Kagoshima-ken
  - Sendai, Kagoshima-ken
  - Shibushi, Kagoshima-ken
  - Soh, Kagoshima-ken
  - So, Kagoshima-ken
  - Tsuruda, Kagoshima-ken
  - Ashigarashimo, Kanagawa
  - Atsugi, Kanagawa
  - Chigasaki, Kanagawa
  - Ebina, Kanagawa
  - Fujisawa, Kanagawa
  - Hiratsuka, Kanagawa
  - Isehara, Kanagawa
  - Kamakura, Kanagawa
  - Kawasaki, Kanagawa
  - Miura, Kanagawa
  - Naka, Kanagawa
  - Odawara, Kanagawa
  - Sagamihara, Kanagawa
  - Yamato, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Zama, Kanagawa
  - Aki, Kochi
  - Muroto, Kochi
  - Nagaoka, Kochi
  - Nankoku, Kochi
  - Takaoka, Kochi
  - Amakusa, Kumamoto
  - Arao, Kumamoto
  - Aso, Kumamoto
  - Hitoyoshi, Kumamoto
  - Kamiamakusa, Kumamoto
  - Kamimashiki, Kumamoto
  - Kōshi, Kumamoto
  - Minamata, Kumamoto
  - Tamana, Kumamoto
  - Uki, Kumamoto
  - Yamaga, Kumamoto
  - Yatsushiro, Kumamoto
  - Fukuchiyama, Kyoto
  - Jōyō, Kyoto
  - Kameoka, Kyoto
  - Kizugawa, Kyoto
  - Kōtari, Kyoto
  - Kyōtanabe, Kyoto
  - Maizuru, Kyoto
  - Nantan, Kyoto
  - Soraku, Kyoto
  - Tsuzuki, Kyoto
  - Uji, Kyoto
  - Yosa, Kyoto
  - Iga, Mie-ken
  - Ise, Mie-ken
  - Kameyama, Mie-ken
  - Kumano, Mie-ken
  - Kuwana, Mie-ken
  - Matsusaka, Mie-ken
  - Suzuka, Mie-ken
  - Tamaru, Mie-ken
  - Tsu, Mie-ken
  - Yokkaichi, Mie-ken
  - Ishinomaki, Miyagi
  - Iwanuma, Miyagi
  - Kesennuma, Miyagi
  - Kurihara, Miyagi
  - Kurokawa, Miyagi
  - Murata, Miyagi
  - Natori-shi, Miyagi
  - Oshika, Miyagi
  - Ōsaki, Miyagi
  - Sendai, Miyagi
  - Shiogama, Miyagi
  - Toda, Miyagi
  - Tome, Miyagi
  - Higashimorokata, Miyazaki
  - Hyūga, Miyazaki
  - Kobayashi, Miyazaki
  - Koyu, Miyazaki
  - Kushima, Miyazaki
  - Miyakonojō, Miyazaki
  - Nichinan, Miyazaki
  - Nishiusuki, Miyazaki
  - Nobeoka, Miyazaki
  - Saito, Miyazaki
  - Azumino, Nagano
  - Chikuma, Nagano
  - Chino, Nagano
  - Hanishina, Nagano
  - Higashichikuma, Nagano
  - Iida, Nagano
  - Ina, Nagano
  - Kamiminochi, Nagano
  - Kiso, Nagano
  - Kitaazumi, Nagano
  - Kitasaku, Nagano
  - Komagane, Nagano
  - Komoro, Nagano
  - Matsumoto, Nagano
  - Okaya, Nagano
  - Saku, Nagano
  - Shimoina, Nagano
  - Shiojiri, Nagano
  - Suwa, Nagano
  - Suzaka, Nagano
  - Ueda, Nagano
  - Gotō, Nagasaki
  - Isahaya, Nagasaki
  - Kitamatsuura, Nagasaki
  - Minamishimabara, Nagasaki
  - Nishisonogi, Nagasaki
  - Ōmura, Nagasaki
  - Sasebo, Nagasaki
  - Shimabara, Nagasaki
  - Sonogishukugō, Nagasaki
  - Tsushima, Nagasaki
  - Unzen, Nagasaki
  - Gose, Nara
  - Ikoma, Nara
  - Kashiba, Nara
  - Kashihara, Nara
  - Kitakatsuragi, Nara
  - Ōuda-yamaguchi, Nara
  - Sakurai, Nara
  - Tenri, Nara
  - Yamatokōriyama, Nara
  - Yamatotakada, Nara
  - Yoshinoyama, Nara
  - Gosen, Niigata
  - Jōetsu, Niigata
  - Kashiwazaki, Niigata
  - Minamiuonuma, Niigata
  - Mitsuke, Niigata
  - Murakami, Niigata
  - Nagaoka, Niigata
  - Ojiya, Niigata
  - Sado, Niigata
  - Sanjō, Niigata
  - Shibata, Niigata
  - Uonuma, Niigata
  - Hita, Oita Prefecture
  - Kunisaki, Oita Prefecture
  - Nakatsu, Oita Prefecture
  - Saiki, Oita Prefecture
  - Tsukawaki, Oita Prefecture
  - Tsukumiura, Oita Prefecture
  - Usa, Oita Prefecture
  - Usuki, Oita Prefecture
  - Yufu, Oita Prefecture
  - Akaiwa, Okayama-ken
  - Asakuchi, Okayama-ken
  - Bizen, Okayama-ken
  - Kaga, Okayama-ken
  - Kasaoka, Okayama-ken
  - Kume, Okayama-ken
  - Kurashiki, Okayama-ken
  - Mimasaka, Okayama-ken
  - Niimi, Okayama-ken
  - Sōja, Okayama-ken
  - Takahashi, Okayama-ken
  - Tamano, Okayama-ken
  - Tomata, Okayama-ken
  - Tsuyama, Okayama-ken
  - Ginowan, Okinawa
  - Ishigaki, Okinawa
  - Itoman, Okinawa
  - Kunigami, Okinawa
  - Miyakojima, Okinawa
  - Naha, Okinawa
  - Nakagami, Okinawa
  - Nanjō, Okinawa
  - Tomigusuku, Okinawa
  - Urasoe, Okinawa
  - Uruma, Okinawa
  - Daitō, Osaka
  - Fujiidera, Osaka
  - Habikino, Osaka
  - Hannan, Osaka
  - Higashiosaka, Osaka
  - Hirakata, Osaka
  - Ibaraki, Osaka
  - Ikeda, Osaka
  - Izumi, Osaka
  - Izumiōtsu, Osaka
  - Izumisano, Osaka
  - Kadoma, Osaka
  - Kaizuka, Osaka
  - Kashihara, Osaka
  - Katano, Osaka
  - Kawachi-Nagano, Osaka
  - Kishiwada, Osaka
  - Matsubara, Osaka
  - Mino, Osaka
  - Moriguchi, Osaka
  - Neyagawa, Osaka
  - Sakai, Osaka
  - Sayama, Osaka
  - Sennan, Osaka
  - Settsu, Osaka
  - Suita, Osaka
  - Takaishi, Osaka
  - Takatsuki, Osaka
  - Tondabayashi, Osaka
  - Toyonaka, Osaka
  - Yao, Osaka
  - Yono, Osaka
  - Imari, Saga-ken
  - Kanzaki, Saga-ken
  - Karatsu, Saga-ken
  - Kishima, Saga-ken
  - Nishimatsuura, Saga-ken
  - Ogi, Saga-ken
  - Takeo, Saga-ken
  - Taku, Saga-ken
  - Tosu, Saga-ken
  - Ureshino, Saga-ken
  - Ageo, Saitama
  - Asaka, Saitama
  - Chichibu, Saitama
  - Fujimi, Saitama
  - Fujimino, Saitama
  - Fukaya, Saitama
  - Gyōda, Saitama
  - Hannō, Saitama
  - Hanyū, Saitama
  - Hasuda, Saitama
  - Hidaka, Saitama
  - Hiki, Saitama
  - Honjō, Saitama
  - Iruma, Saitama
  - Kasukabe, Saitama
  - Kawagoe, Saitama
  - Kawaguchi, Saitama
  - Kazo, Saitama
  - Kitaadachi, Saitama
  - Kitamoto, Saitama
  - Koshigaya, Saitama
  - Kōnosu, Saitama
  - Kukichūō, Saitama
  - Kumagaya, Saitama
  - Minamisaitama, Saitama
  - Niiza, Saitama
  - Sakado, Saitama
  - Sayama, Saitama
  - Sōka, Saitama
  - Toda, Saitama
  - Tokorozawa, Saitama
  - Tsurugashima, Saitama
  - Wako, Saitama
  - Yoshikawa, Saitama
  - Higashiōmi, Shiga
  - Hikone, Shiga
  - Inukami, Shiga
  - Kōka, Shiga
  - Kusatsu, Shiga
  - Moriyama, Shiga
  - Nagahama, Shiga
  - Ōmihachiman, Shiga
  - Ōtsu, Shiga
  - Rittō, Shiga
  - Takashima, Shiga
  - Hamada, Shimane
  - Izumo, Shimane
  - Kanoashi, Shimane
  - Matsue, Shimane
  - Nita, Shimane
  - Oda, Shimane
  - Unnan, Shimane
  - Yasugi, Shimane
  - Atami, Shizuoka
  - Fuji, Shizuoka
  - Fujieda, Shizuoka
  - Fujinomiya, Shizuoka
  - Fukuroi, Shizuoka
  - Gotemba, Shizuoka
  - Haibara, Shizuoka
  - Hamamatsu, Shizuoka
  - Itō, Shizuoka
  - Iwata, Shizuoka
  - Izu, Shizuoka
  - Kakegawa, Shizuoka
  - Kamo, Shizuoka
  - Kikugawa, Shizuoka
  - Kosai, Shizuoka
  - Mishima, Shizuoka
  - Numazu, Shizuoka
  - Omaezaki, Shizuoka
  - Shimada, Shizuoka
  - Shimoda, Shizuoka
  - Susono, Shizuoka
  - Tagata, Shizuoka
  - Ashikaga, Tochigi
  - Kanuma, Tochigi
  - Kawachi, Tochigi
  - Mooka, Tochigi
  - Nasu, Tochigi
  - Nasukarasuyama, Tochigi
  - Nikkō, Tochigi
  - Oyama, Tochigi
  - Ōtawara, Tochigi
  - Sano, Tochigi
  - Ubagai, Tochigi
  - Utsunomiya, Tochigi
  - Anan, Tokushima
  - Awa, Tokushima
  - Mima, Tokushima
  - Miyoshi, Tokushima
  - Myozai, Tokushima
  - Naka, Tokushima
  - Narutochō-mitsuishi, Tokushima
  - Okuno, Tokushima
  - Yoshinogawa, Tokushima
  - Adachi City, Tokyo
  - Akiruno, Tokyo
  - Akishima, Tokyo
  - Arakawa City, Tokyo
  - Bunkyo, Tokyo
  - Chiyoda City, Tokyo
  - Chōfu, Tokyo
  - Chūō, Tokyo
  - Edogawa City, Tokyo
  - Fuchū, Tokyo
  - Fussa, Tokyo
  - Hachiōji, Tokyo
  - Higashiyamato, Tokyo
  - Hino, Tokyo
  - Inagi, Tokyo
  - Katsushika-ku, Tokyo
  - Kita-ku, Tokyo
  - Kiyose, Tokyo
  - Kodaira, Tokyo
  - Koganei, Tokyo
  - Kokubunji, Tokyo
  - Komae, Tokyo
  - Koto, Tokyo
  - Kunitachi, Tokyo
  - Machida, Tokyo
  - Meguro City, Tokyo
  - Minato, Tokyo
  - Mitaka, Tokyo
  - Musashino, Tokyo
  - Nakano City, Tokyo
  - Nerima City, Tokyo
  - Nishitōkyō, Tokyo
  - Ōme, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya City, Tokyo
  - Shibuya City, Tokyo
  - Shinagawa, Tokyo
  - Shinjuku, Tokyo
  - Suginami, Tokyo
  - Sumida City, Tokyo
  - tabashi City, Tokyo
  - Tachikawa, Tokyo
  - Tama, Tokyo
  - Toshima City, Tokyo
  - Iwai, Tottori
  - Kōge, Tottori
  - Kurayoshi, Tottori
  - Neu, Tottori
  - Saihaku, Tottori
  - Sakaiminato, Tottori
  - Yonago, Tottori
  - Himi, Toyama
  - Imizu, Toyama
  - Nakaniikawa, Toyama
  - Namerikawa, Toyama
  - Nanto, Toyama
  - Takaoka, Toyama
  - Uozu, Toyama
  - Arida, Wakayama
  - Gobō, Wakayama
  - Ito, Wakayama
  - Iwade, Wakayama
  - Kainan, Wakayama
  - Kinokawa, Wakayama
  - Nishimuro, Wakayama
  - Tanabe, Wakayama
  - Nanyō, Yamagata
  - Sakata, Yamagata
  - Tendō, Yamagata
  - Tsuruoka, Yamagata
  - Yonezawa, Yamagata
  - Hagi, Yamaguchi
  - Hikari, Yamaguchi
  - Hōfu, Yamaguchi
  - Iwakuni, Yamaguchi
  - Nagato, Yamaguchi
  - Sanyōonoda, Yamaguchi
  - Shimonoseki, Yamaguchi
  - Shūnan, Yamaguchi
  - Ube, Yamaguchi
  - Yanai, Yamaguchi
  - Chūō, Yamanashi
  - Fuefuki, Yamanashi
  - Fujiyoshida, Yamanashi
  - Hokuto, Yamanashi
  - Kai, Yamanashi
  - Kofu, Yamanashi
  - Minamitsuru, Yamanashi
  - Nirasaki, Yamanashi
  - Ōtsuki, Yamanashi
  - Tsuru, Yamanashi
  - Aichi
  - Akita
  - Aomori
  - Chiba
  - Fukui
  - Fukuoka
  - Fukushima
  - Gifu
  - Hiroshima
  - Ishikawa
  - Kagoshima
  - Kochi
  - Kumamoto
  - Kyoto
  - Mie
  - Miyagi
  - Miyazaki
  - Nagano
  - Nagasaki
  - Nara
  - Niigata
  - Okayama
  - Okinawa
  - Osaka
  - Ōita
  - Saga
  - Saitama
  - Shizuoka
  - Tochigi
  - Tokushima
  - Tottori
  - Toyama
  - Wakayama
  - Yamagata
  - Yamaguchi

REFERENCES:
- [Background] Arai H, Hashimoto N, Sumitomo K, Takase T, Ishii M. Disease state changes and safety of long-term donepezil hydrochloride administration in patients with Alzheimer's disease: Japan-Great Outcome of Long-term trial with Donepezil (J-GOLD). Psychogeriatrics. 2018 Sep;18(5):402-411. doi: 10.1111/psyg.12340. Epub 2018 Jul 11. PMID 29993162